CLINICAL TRIAL: NCT07043400
Title: A Phase 3, Multi-Center, Randomized, Open-Label Clinical Study of Tislelizumab Administered as Subcutaneous Injection Versus Intravenous Infusion Plus Chemotherapy as First-Line Treatment in Patients With Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: A Study to Investigate Tislelizumab Administered as Subcutaneous Injection Versus Intravenous Infusion Plus Chemotherapy in Patients With Unresectable or Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-316; 2025-522862-58-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — tislelizumab; Cisplatin; Leucovorin; Fluorouracil; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Tislelizumab Subcutaneous + Chemotherapy (Experimental): Participants will receive tislelizumab 300 mg subcutaneous (SC) injection on Day 1 of each 21-day cycle, followed by chemotherapy decided on an individual patient basis.
  Interventions: Drug: Subcutaneous Tislelizumab; Drug: Cisplatin; Drug: Leucovorin; Drug: 5-fluorouracil (5-FU); Drug: Oxaliplatin; Drug: Capecitabine
- Arm B: Tislelizumab Intravenous Infusion + Chemotherapy (Active Comparator): Participants will receive tislelizumab 200 mg intravenous infusion (IV) on Day 1 of each 21-day cycle, followed by chemotherapy decided on an individual patient basis.
  Interventions: Drug: Intravenous Tislelizumab; Drug: Cisplatin; Drug: Leucovorin; Drug: 5-fluorouracil (5-FU); Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Subcutaneous Tislelizumab — Administered by subcutaneous injection
  Other Names: BGB-A317
  Arms: Arm A: Tislelizumab Subcutaneous + Chemotherapy
Drug: Intravenous Tislelizumab — Administered by intravenous infusion
  Other Names: BGB-A317; TEVIMBRA®
  Arms: Arm B: Tislelizumab Intravenous Infusion + Chemotherapy
Drug: Cisplatin — Administered by intravenous infusion
Drug: Leucovorin — Administered by intravenous infusion
Drug: 5-fluorouracil (5-FU) — Administered by intravenous infusion
Drug: Oxaliplatin — Administered by intravenous infusion
Drug: Capecitabine — Administered orally

SUMMARY:
This study is designed to assess the levels of drug exposure following treatment with tislelizumab administered as a subcutaneous (SC) injection compared to intravenous infusion (IV) as first-line therapy in adults with gastric or gastroesophageal junction (GEJ) that is locally advanced and cannot be surgically removed or has spread from the stomach to other areas of the body. Approximately 351 patients will be participating in this study. The study is composed of a screening period, a treatment period, and a follow-up period.

DETAILED DESCRIPTION:
Our company, previously known as BeiGene, is now officially BeOne Medicines. Because some of our older studies were sponsored under the name BeiGene, you may see both names used for this study on this website.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced unresectable or metastatic gastric/ gastroesophageal junction (GEJ) adenocarcinoma.
* No previous systemic therapy for locally advanced unresectable or metastatic gastric/GEJ cancer.
* At least 1 measurable or nonmeasurable lesion per RECIST v1.1 as determined by investigator assessment.
* Must be able to provide tumor tissues for biomarker assessment.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score ≤ 1.
* Adequate organ function.
* Women of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study and ≥ 120 days after the last dose of tislelizumab.
* Non-sterile males must be willing to use a highly effective method of birth control for the duration of the study and for ≥ 120 days after the last dose of tislelizumab.

Exclusion Criteria:

* Squamous cell or undifferentiated or other histological type gastric cancer (GC)
* Active leptomeningeal disease or uncontrolled brain metastasis. Patients with equivocal findings or with confirmed brain metastases are eligible for enrollment provided that they are asymptomatic and radiologically stable without the need for corticosteroid treatment for ≥ 4 weeks before randomization.
* Diagnosis with gastric or GEJ adenocarcinoma with positive human epidermal growth factor receptor 2 (HER2).
* Active autoimmune diseases or history of autoimmune diseases that may relapse.
* Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (at least once a week) and/or diuretics within 7 days prior to randomization

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-04-22 (Estimated)

PRIMARY OUTCOMES:
Model-Predicted Steady State Trough Concentration (Ctrough) of Tislelizumab | 85 Days
Model-Predicted Area under the Concentration-time Curve from Time Zero to 21 Days (AUC0-21d) after the First Dose of Tislelizumab | 21 Days

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of participants with partial or complete response, as assessed by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from randomization date until first documentation of progression or death, whichever comes first, as assessed by the investigator using RECIST v1.1
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from the date that response criteria are first met to the date that progressive disease is objectively documented or death, whichever comes first as assessed by the investigator using RECIST v1.1
Disease Control Rate (DCR) | Up to 2 years
  DCR is defined as the percentage of participants whose best overall response is complete response, partial response, or stable disease, as assessed by the investigator using RECIST v1.1
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from first study drug administration to the date of death due to any cause
Number of Participants With Adverse Events (AEs) | Up to 2 years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory values, vital signs, physical examination findings, and electrocardiogram results.
Model-predicted Serum Ctrough at Cycle 1 | 21 Days
Observed Serum Ctrough at Cycle 1 | 21 Days
Observed Area Under the Concentration-time Curve at Steady-state (AUC) at Cycle 1 | 21 Days
Model-predicted Area Under the Concentration-time Curve at Steady-state (AUCss) | 85 Days
Percentage of Participants with Antidrug Antibodies (ADAs) to Tislelizumab after SC or IV Administration | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (65):
- United States (15):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - Bioresearch Partners Holding Hialeah Hospital, Hialeah, Florida
  - Orlando Health Ufhealth Cancer Center, Orlando, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - New England Cancer Specialists, Westbrook, Maine
  - St Louis Cancer Care, Llp, Bridgeton, Missouri
  - Nebraska Hematology Oncology, Lincoln, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - Oregon Oncology Specialists, Salem, Oregon
  - Md Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties, Tacoma, Washington
- Brazil (10):
  - Hospital de Amor Barretos, Barretos
  - CECAP, Blumenau
  - Hospital Brasilia, Brasília
  - Hospital Sao Lucas Da Pucrs, Porto Alegre
  - IMIP, Recife
  - Inca Instituto Nacional de Cancer, Rio de Janeiro
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto
  - Icesp Instituto Do Cancer Do Estado de Sao Paulo Octavio Frias de Oliveira, São Paulo
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Hospital Santa Rita de Cassia Afecc, Vitória
- China (15):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Anyang Tumor Hospital, Anyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Nanjing Drum Tower Hospital,the Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Ganzhou Peoples Hospital Ganzhou Hospital Affiliated to Nanchang University, Ganzhou, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Changzhi Peoples Hospital, Changzhi, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Czechia (3):
  - Masarykuv Onkologicky Ustav, Brno
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Olomouc, Olomouc
- France (2):
  - Institut Sainte Catherine, Avignon
  - Chru de Brest Hopital Cavale Blanche, Brest
- Japan (8):
  - Japan Community Health Care Organization Kyushu Hospital, Kitakyushu, Fukuoka
  - Nho Hokkaido Cancer Center, Sapporo, Hokkaido
  - Osaka Rosai Hospital, SakaiShi, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsukishi, Osaka
  - Saitama Cancer Center, Kitaadachigun, Saitama
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Institute of Science Tokyo Hospital, Bunkyoku, Tokyo
  - Tokyo Metropolitan Bokutoh Hospital, SumidaKu, Tokyo
- Pan American Oncology Trials, Llc, Rio Piedras, Puerto Rico
- South Korea (6):
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, BukGu, Gyeongsangbukdo
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Ninewells Hospital and Medical School, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/